CLINICAL TRIAL: NCT04543513
Title: Self-regulation of Prefrontal Cortex During Emotional Cognitive Control in PTSD
Acronym: SPrC-PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes to protocol are necessary to optimize engagement of neural target
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Principal Investigator, Robin Aupperle, Principal Investigator, Laureate Institute for Brain Research, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-012 - Part 2
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: PTSD; Cognitive Function
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Left Dorsolateral Prefrontal Cortex rtfMRI-nf (Experimental): Real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) will target left dorsolateral prefrontal cortex. Participants in this arm will receive active feedback while attempting to modulate their neural activity during an emotional cognitive control task.
  Interventions: Other: Real-time functional magnetic resonance neurofeedback (rtfMRI-nf)

INTERVENTIONS:
Other: Real-time functional magnetic resonance neurofeedback (rtfMRI-nf) — Real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) is a procedure using an MRI scanner that allows participants to observe their own neural activity in the moment. They are taught to self-regulate this activity during a task.

SUMMARY:
Deficits in emotional cognitive control are present in a number of clinical psychiatric populations including depression, anxiety, and PTSD. Deficits in this domain of function limit one's ability to focus attention on goal-directed activities while inhibiting reactions to irrelevant emotional stimuli, and this contributes to the symptoms of these disorders and makes individuals less likely to be successful in existing treatments. The left dorsolateral prefrontal cortex (LDLPFC) and its connectivity with other regions (i.e., dorsal anterior cingulate cortex, ventromedial prefrontal cortex, insula, amygdala) is thought to play a central role in facilitating emotional cognitive control. However, past research has primarily utilized correlational approaches that limit conclusions about the directionality of these relationships. Enhancing our understanding of the neural underpinnings of emotional cognitive control could be valuable for informing treatment for populations with deficits in these processes, such as adults with PTSD.

The current study utilizes a neuromodulatory approach called real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) whereby participants observe their own neural activity in the moment and are taught to self-regulate this activity. Adult volunteers, who have been diagnosed with PTSD, will be trained to increase neural activity in LDLPFC while involved in mental tasks involving emotional cognitive control processes. The mental tasks will include counting, remembering words, or planning events while viewing negatively-valenced emotional words (e.g., kill, death, threat). Participants in this study will complete a non-randomized LDLPFC rtfMRI-nf protocol to assess tolerability and feasibility of the protocol in a clinical population of interest. Resting-state fMRI scans and behavioral testing sessions will take place before and after rtfMRI-nf.

The specific aims are to examine the impact of LDLPFC rtfMRI-nf on: (1) LDLPFC activity during emotional cognitive control, (2) LDLPFC functional connectivity with other brain regions during rest, and (3) cognitive control task performance. As this study is meant to be preliminary, the target sample size is not powered to detect statistical significance for these measures. However, effect size estimates will be calculated to provide potential justification for future work with this protocol in this clinical population.

To these ends, this study will use rtfMRI-nf to examine preliminary evidence of a novel protocol to regulate LDLPFC activity in adults diagnosed with PTSD. This research will improve our understanding of emotional cognitive control and demonstrate whether this is a modifiable target for intervention in this clinical population of interest.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* sufficient English proficiency to complete procedures
* primary DSM-5 psychiatric diagnosis of posttraumatic stress disorder (PTSD)

Exclusion Criteria:

* significant or unstable physical or mental health conditions (e.g., immediate suicidal intent) requiring medical attention
* meeting criteria in either the present or past for the following DSM-5 psychiatric disorders: Schizophrenia Spectrum and Other Psychotic Disorders, Obsessive- Compulsive disorders, or Bipolar and Related Disorders
* recent change (i.e., within 6 weeks) for prescription of psychiatric medication
* current, regular benzodiazepine use
* history of moderate to severe traumatic brain injury
* diagnosis of neurologic disorders
* current alcohol/drug abuse
* MRI contra-indications (e.g., metal in body)
* uncorrected vision/hearing problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Left dorsolateral prefrontal cortex activity during emotional cognitive control (pre- to post-neurofeedback) | Approximately 2 hours after baseline assessment
  Individual ability to regulate left dorsolateral prefrontal cortex activity during an emotional cognitive control task will be assessed before and after neurofeedback.

SECONDARY OUTCOMES:
Left dorsolateral prefrontal cortex functional connectivity with other brain regions during rest (pre- to post-neurofeedback) | Approximately 2 hours after baseline assessment
  Individual functional connectivity values between left dorsolateral prefrontal cortex and other brain regions during rest will be assessed before and after neurofeedback.

OTHER OUTCOMES:
Emotional Stroop Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the emotion condition of the emotional Stroop task.
Color Word Stroop Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the inhibition condition of the color word Stroop task.
Flanker Task Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the incongruent condition of the Flanker task.
Emotional Stroop Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for emotional versus neutral conditions of the emotional Stroop task.
Color Word Stroop Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for inhibition versus reading conditions of the emotional Stroop task.
Flanker task Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for incongruent versus congruent conditions of the Flanker task.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Aupperle, Ph.D., Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be released publicly, but requests for group-averaged results will be considered by individual request following publication of findings from this study.